CLINICAL TRIAL: NCT04223492
Title: Liquid Biopsies and Imaging in Breast Cancer
Acronym: LIMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Horizon 2020 - European Commission (Other); Philips Electronics Nederland BV (Industry); Agena Bioscience GmbH (Unknown); DiaDx (Unknown); Stilla Technologies (Unknown); ANGLE Europe Limited (Unknown); ALS Automated Lab Solutions GmbH (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Philips GmbH Innovate Technologies (Unknown); Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Principal Investigator, Dr. Kenneth Gilhuijs, Associate Professor, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-396
Record Dates: First submitted 2019-12-20; First posted 2020-01-10 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Neoadjuvant; Response Prediction; Liquid Biopsies; Magnetic resonance imaging; Circulating Tumor DNA
MeSH Terms: conditions — Breast Neoplasms | interventions — Liquid Biopsy; Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant systemic treatment (Other): All patients undergo standard neoadjuvant treatment and additional multi-parametric MRI and liquid biopsies during neoadjuvant treatment.
  Interventions: Diagnostic Test: Liquid biopsy; Diagnostic Test: Multi-parametric MRI

INTERVENTIONS:
Diagnostic Test: Liquid biopsy — A blood sample containing circulating tumor DNA and circulating tumor cells.
Diagnostic Test: Multi-parametric MRI — Multi-parametric MRI combines different imaging protocols in one session to measure more functional items than perfusion alone, addressing different aspects of tumor biology.

SUMMARY:
The aim of the study is to show proof of concept for combining multi-parametric MRI with liquid biopsies in addition to conventional clinical and pathologic information, to accurately predict response to neoadjuvant treatment for patients with primary breast cancer.

DETAILED DESCRIPTION:
The response to neoadjuvant chemotherapy (NAC) in early stage breast cancer has important prognostic implications. Early, dynamic prediction of response allows for adaption of the treatment plan before completion, or even before the start of treatment. This strategy can help prevent overtreatment and related toxicity and correct for undertreatment with an ineffective regimen. The hypothesis of this study is that accurate dynamic response prediction may be reached by combining multi-parametric MRI with liquid biopsies prior to, during and after NAC, in addition to conventional clinical and pathological information. Magnetic resonance imaging (MRI) is non-invasive and is typically used for response evaluation in current clinical practice. It shows the size and perfusion of the tumor as they change during treatment. However, tumor size on MRI has limited predictive value for response to therapy. Multi-parametric MRI uses different imaging protocols in one session to measure more functional items than perfusion alone, addressing different aspects of tumor biology, and possibly improving predictive value. With this improvement, imaging still only visualizes macroscopic disease. Therefore, in the LIMA study, MRI will be combined with liquid biopsies containing circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA), which have both shown prognostic and predictive values in early stage breast cancer. Since the ctDNA may originate from cells in every part of the tumor, it may capture tumor heterogeneity. Liquid biopsies are minimally invasive and provide insight into microscopic tumor load and the tumor's genetic picture.

The aim of the study is to show proof of concept for combining multi-parametric MRI with liquid biopsies in addition to conventional clinical and pathologic information, to accurately predict response to neoadjuvant treatment for patients with primary breast cancer.

The LIMA is a multicenter prospective observational cohort study. Multi-parametric MRI will we performed prior to NAC, halfway and after completion of NAC. Liquid biopsies will be obtained before start of treatment, every 2 weeks during treatment and after completion of NAC. 100 patients will be enrolled in different hospitals.

Funding from the European Union Horizon 2020 research and innovation program under grant agreement no. 755333 (LIMA)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive breast carcinoma
* Planned for neoadjuvant chemotherapy (and in case of a Her2-positive tumor: addition of trastuzumab and/or pertuzumab)

Exclusion Criteria:

* Luminal A breast cancer (defined as: ER-positive and HER2-negative by immunohistochemistry and Bloom and Richardson grade 1 or 2)
* Inflammatory breast cancer
* Distant metastases on PET/CT
* Other active malignant disease in the past 5 years (excluded squamous cell or basal cell carcinoma of the skin)
* Pregnant or lactating women
* Contra-indications for MRI according to standard hospital guidelines
* Contra-indications for gadolinium-based contrast-agent, including known prior allergic reaction to any contrast-agent, and renal failure, defined by GFR < 30 mL/min/1.73m2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Residual Cancer Burden index in surgical resection specimen | After neoadjuvant treatment and surgery (approx. 6 months from diagnosis)
  The following parameters are required from pathologic examination in order to calculate Residual Cancer Burden (RCB) after neoadjuvant treatment: Primary tumor bed area, overall cancer cellularity (as percentage of area), percentage of cancer that is in situ disease, number of positive lymph nodes and diameter of largest metastasis. These parameters are filled in in the calculator that is available online to calculate the Residual Cancer Burden index: http://www3.mdanderson.org/app/medcalc/index.cfm?pagename=jsconvert3

SECONDARY OUTCOMES:
Radiological lesion volume on DCE MRI after NAC | After neoadjuvant treatment (approx. 6 months from diagnosis)
  Measured in three dimensions as described in ACR BI-RADS Atlas® 5th Edition
pathological complete response, defined as ypT0/ypN0 | After neoadjuvant treatment and surgery (approx. 6 months from diagnosis)
  Pathological complete response, defined as ypT0/ypN0

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth GA Gilhuijs, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Meta-data will be made publicly available. A steering committee will assess any request for reuse of the data.
Supporting Information: Study Protocol, SAP
Time Frame: Within 2 years after the LIMA Project has ended (and the LIMA breast cancer trial thus has been closed by the IRB)
Access Criteria: Any reasonable request compliant with patient consent will be granted.

REFERENCES:
- [Derived] Janssen LM, Suelmann BBM, Elias SG, Janse MHA, van Diest PJ, van der Wall E, Gilhuijs KGA. Improving prediction of response to neoadjuvant treatment in patients with breast cancer by combining liquid biopsies with multiparametric MRI: protocol of the LIMA study - a multicentre prospective observational cohort study. BMJ Open. 2022 Sep 20;12(9):e061334. doi: 10.1136/bmjopen-2022-061334. PMID 36127090